CLINICAL TRIAL: NCT06835660
Title: DRug-Eluting BallOOn Versus Primary Polymer-coated Paclitaxel Eluting STenting for Femoro-popliteal Lesions
Acronym: REBOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24RCS-REBOOST
Record Dates: First submitted 2025-02-10; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Femoropopliteal Lesion
Keywords: femoropopliteal lesion; lower limb peripheral arterial disease; self-expandable bare metal stent; plain balloon angioplasty; self expandable polymer-coated paclitaxel eluting stents; drug-coated balloon

STUDY DESIGN:
Who Masked: Participant
Masking Description: This is a single blind study. Patients will not be aware of the treatment received at the level of the FPL (DCB or SEBMS). During the procedure and the duplex-scan examinations for follow-up, the medical team will not use any term allowing the patient to know which medical device is used. The operative and the duplex-scan reports will not allow to know in the which treatment arm is the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (DCB) (Active Comparator): Drug coated balloon(s) will be used for femoropopliteal lesions.
  Patients assigned to the DCB group (study group) will receive DCB inflation(s) at the level of the lesions according the DCB instructions for use.
  Interventions: Device: procedure of DCB implantation
- Comparator group (SEBMS) (Active Comparator): Uncovered self-expandable polymer coated paclitaxel eluting stent(s) will be used for femoropopliteal lesions.
  Patients assigned to the SEDES group (control group) will receive implantation ELUVIA stents at the level of the lesion(s) according to the SEDES instructions for use.
  Interventions: Device: procedure of SEDES implantation

INTERVENTIONS:
Device: procedure of DCB implantation — Patients assigned to the DCB group (study group) will receive DCB inflation(s) at the level of the lesions according the DCB instructions for use (120 seconds inflation minimum). One or several DCBs will be inflated at the level of the lesions depending on lesions' lengths. The DCB diameter(s) will be the one(s) of the index diameter of the artery. Overlaps between zones that will receive DCB inflations will be of 10 mm to avoid any geographic miss.
  Arms: Study group (DCB)
Device: procedure of SEDES implantation — SEDES implantation wille be performed according to the SEDES instructions for use. Stent(s) oversizing will be of 1 mm maximum. Overlaps between stents will be of 10 mm.
  Completion angiogram will assess the technical success of the procedure (see endpoints definitions). The physician may then decide to add a bailout SEBMS because of flow limiting dissection and/or a new stenosis >30%.
  Arms: Comparator group (SEBMS)

SUMMARY:
Main objective of the study: To demonstrate that a primary DCB strategy is non-inferior in terms of primary patency to a primary SEDES strategy for above-the-knee femoro-popliteal lesions at 12 months.

Primary endpoint: Freedom from loss of primary patency at 12 months: loss of primary patency will be defined as the need for target vessel revascularization and/or binary restenosis (defined as >70% in diameter or peak systolic velocity >2.4 m/sec at duplex examination).

Secondary objectives:

To demonstrate that a primary DCB strategy is non-inferior to a primary SEDES strategy in terms of:

* Intra-operative technical success.
* Safety at 1, 6, 12, 18 and 24 months.
* Primary patency at 1, 6, 12, 18 and 24 months.
* Assisted primary patency at 1, 6, 12, 18 and 24 months.
* Secondary patency at 1, 6, 12, 18 and 24 months.
* All target vessel revascularization at 1, 6, 12, 18 and 24 months.
* Clinically-driven target vessel revascularization at 1, 6, 12, 18 and 24 months.
* All TLR at 1, 6, 12, 18 and 24 months.
* Clinically-driven TLR at 1, 6, 12, 18 and 24 months.
* All target extremity revascularization at 1, 6, 12, 18 and 24 months.
* Number of secondary interventions at 1, 6, 12, 18 and 24 months.
* Binary restenosis at 1, 6, 12, 18 and 24 months.
* Mean Rutherford category at 1, 6, 12, 18 and 24 months.
* Mean ABI value at 1, 6, 12, 18 and 24 months.
* Absolute claudication distance improvement at 1, 6, 12, 18 and 24 months.
* Quality of life at 1, 6, 12, 18 and 24 months.
* Cost at 1, 6, 12, 18 and 24 months.

DETAILED DESCRIPTION:
Femoropopliteal lesions (FPL) are the most common localization of lower limb peripheral arterial disease (LLPAD). Previous prospective randomized studies conducted in the 2000s demonstrated the superiority of self-expandable bare metal stent (SEBMS) placement over plain balloon angioplasty (PBA) in FPL at 12 months, 24 months and beyond. Recent studies show a significant benefit of self expandable polymer-coated paclitaxel eluting stents (SEDES) over SEBMS and led to consider SEDES implantation as the treatment of choice for FPL, especially in France with ≈45 000 self expandable stents implantations per year at this level. More recently, prospective randomized trials demonstrated that drug-coated balloon (DCB) use was superior to PBA in FPL at 12 months, 24 months and beyond. Primary patency at 12 months of both SEDES and DCB appeared in the same ranges.

SEDES and DCB are therefore now recognized as two valuable options for FPL and they are both reimbursed for the treatment of such lesions. However, the choice between the two treatment strategies remains unclear. On one hand, primary SEDES allows a secure approach that limits the risk of post-angioplasty dissection and thrombosis, but a permanent metallic scaffold remains inside the treated artery, with a late risk of stent fracture and challenging in-stent restenosis. On the other hand, DCB may be at risk of early arterial recoil but allows leaving nothing behind in the arterial bed. Early recoil mandates self expandable stents implantation after DCB with an increased procedural cost in approximately 10% of patients. Since no rigorous independent trial directly compared these two strategies, this study will prospectively compare SEDES and DCB for above-the-knee FPL.

This study is a non-inferiority, prospective, comparative trial. Patients will be screened using clinical and duplex scan examinations. Patients matching inclusion criteria and without exclusion criteria will give written informed consent before the endovascular revascularization procedure.

Technically, following puncture of the femoral artery, an angiogram will be performed. The lesion(s) will be identified and crossed by a guidewire. Vessel preparation (predilatation) will be performed using PBA at the level of the lesion up to the index diameter of the artery (60 seconds minimum). Another angiogram will determine technical success or failure of the predilatation. Predilatation success is defined as the absence of flow limiting dissection and/or residual stenosis >30%. Patients with predilatation failure will receive an adequate treatment (generally a provisional stenting) at the physician's discretion. These patients with predilatation failure will not be randomized and will not be further followed in the study. Patients with predilatation success will then be randomized intraoperatively to a DCB or a SEDES strategy using a dedicated web server with stratification on Center, Rutherford category (2-3/4) and lesion length (short vs. long lesion, as described above). Participants will be distributed between groups at a ratio of (1:1).

After the procedure, patients will be prescribed clopidogrel for 90 days and aspirin for lifelong.

Patients will be assessed at 1, 6, 12, 18 and 24 months follow-up with clinical and duplex-scan examination. An independent core laboratory will examine duplex-scan results.

15 national sites/recruitment centers will be involved in the study targetting 402 patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 18
* Subject has been informed of the nature of the study, agrees to participate, and has signed a Medical Ethics Committee approved consent form.
* Rutherford category 2-4.
* Femoro-popliteal stenosis/occlusion
* Target lesion is below the origin of the profunda femoris and does not exceed the medial femoral epicondyle.
* Patent inflow artery (<30% diameter stenosis).
* Patency of at least one infrapopliteal artery to the ankle (<30% diameter stenosis) in continuity with the native femoropopliteal artery.

Exclusion Criteria:

* Inability to obtain informed consent.
* Life expectancy <24 months.
* Pregnancy or breastfeeding during study period.
* Known clotting disorders.
* Contraindication to antiplatelet therapy or anticoagulants.
* Known hypersensitivity to nitinol or paclitaxel.
* Enrollment into another study.
* Significant iliac or common femoral stenosis (<30% diameter) requiring intervention during the index procedure.
* In-stent restenosis
* Total occlusion non-crossable by a guidewire.
* Acute thrombosis of target vessel
* Prior ipsilateral femoro-popliteal bypass.
* Implantation of a drug-eluting stent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Loss of primary patency | at 12 months
  Freedom from loss of primary patency at 12 months: loss of primary patency will be defined as the need for target vessel revascularization and/or binary restenosis.
  defined as >70% in diameter or peak systolic velocity >2.4 m/sec at duplex examination

SECONDARY OUTCOMES:
Intraoperative technical success | through study completion, an average of 24 months
  Intraoperative technical success, defined as the absence of flow limiting dissection or residual stenosis >30% at the final completion angiogram.
Assisted primary patency | at 1, 6, 12, 18 and 24 months
  Assisted primary patency is defined as vessel patency even when maintained by repeated percutaneous intervention, but prior to complete vessel occlusion.
Secondary patency | at 1, 6, 12, 18 and 24 months
  Secondary patency is defined as vessel patency even when maintained by repeated percutaneous intervention, prior or after complete vessel occlusion.
Target vessel revascularization | at 1, 6, 12, 18 and 24 months
  Target vessel revascularization, defined by any secondary intervention on the ipsilateral femoropopliteal artery above the knee.
Clinically-driven target vessel revascularization | at 1, 6, 12, 18 and 24 months
  Clinically-driven target vessel revascularization
Target lesion revascularization (TLR) | at 1, 6, 12, 18 and 24 months
  Target lesion revascularization (TLR) defined by any secondary intervention on the index lesion.
Clinically-driven TLR | at 1, 6, 12, 18 and 24 months
  Clinically-driven TLR
Target extremity revascularization | at 1, 6, 12, 18 and 24 months
  Target extremity revascularization defined by any revascularization on vascular tree of the ipsilateral limb.
Binary restenosis | at 1, 6, 12, 18 and 24 months
  Binary restenosis, defined as >70% or peak systolic velocity >2.4 m/sec at duplex examination
Rutherford category | at 1, 6, 12, 18 and 24 months
  Rutherford category by Rutherford classification
ABI value | at baseline, 1, 6, 12, 18 and 24 months
  ABI value: ankle-brachial index evaluated by clinical examination
Absolute claudication distance improvement | at 1, 6, 12, 18 and 24 months
  Absolute claudication distance improvement: evaluated by clinical interview and examination
Quality of life assessement | at 1, 6, 12, 18 and 24 months
  Quality of life assessed by the Walking Impairment Questionnaire (WIQ)
Cost | at 1, 6, 12, 18 and 24 months
  Cost at 1, 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël COSCAS, MD, PhD, Principal Investigator — Department of Vascular Surgery, Ambroise Paré Hospital - AP-HP
Locations (1):
- Department of Vascular Surgery, Ambroise Paré Hospital - AP-HP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: Undecided